CLINICAL TRIAL: NCT04986046
Title: Fruit and Vegetable Rx + Home Plate, a Multilevel Intervention to Improve Dietary Disparities Among Low-income Children and Families
Brief Title: Fruit and Vegetable Rx (FVRx) + Home Plate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: McClay Foundation (Unknown); University of Pennsylvania (Other); The Leo and Peggy Pierce Family Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-018132
Record Dates: First submitted 2021-06-09; First posted 2021-08-02 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Food Insecurity
Keywords: Diet quality; Cooking; Food security; Food access; Community food environment; Mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fruit and vegetable prescription (Active Comparator): Fruit and vegetable incentive program
  Interventions: Other: Fruit and Vegetable prescription
- Fruit and vegetable prescription + Home Plate Lite (Experimental): Fruit and vegetable incentive program + asynchronous, electronic resources delivered over six weeks (Home Plate Lite)
  Interventions: Other: Home Plate Lite; Other: Fruit and Vegetable prescription
- Fruit and vegetable prescription + Home Plate (Experimental): Fruit and vegetable incentive program + 1.5-hour, virtual, small-group classes weekly for six weeks (Home Plate)
  Interventions: Other: Home Plate; Other: Fruit and Vegetable prescription

INTERVENTIONS:
Other: Home Plate Lite — Home Plate Lite comprises electronic educational content (e.g. recipes, instructional videos) disbursed at least weekly over six weeks.
  Arms: Fruit and vegetable prescription + Home Plate Lite
Other: Home Plate — Home Plate comprises six 1.5-hour weekly sessions where parents work together with a study staff member to discuss the learning objectives and prepare the components of a meal, including entrees, side dishes, and desserts.
  Arms: Fruit and vegetable prescription + Home Plate
Other: Fruit and Vegetable prescription — All families will receive FVRx over two months; FVRx can be redeemed for fresh, frozen, or canned produce at participating retailers in Philadelphia

SUMMARY:
This is a research study to test if fruit and vegetable prescription vouchers (FVRx) and a cooking skills program (Home Plate) can improve dietary quality, food security (access to a sufficient quantity of affordable, nutritious food), feelings about the home and community food environments, and caregiver mental health.

DETAILED DESCRIPTION:
The purpose of this research study is to determine the effect of produce prescriptions (vouchers that can be redeemed for produce at participating locations, "FVRx") and a cooking skills program (Home Plate) on dietary quality, food security, perceptions of the food environment, and mental health. Investigators also aim to determine the feasibility and acceptability of the programs.

ELIGIBILITY:
Inclusion Criteria

1. At least one child in the household is age 2 to 5 years.
2. Household is food insecure and/or low-income with an age-eligible, overweight or obese child.

   * If a child meets the above criteria, any sibling age 2-5 is also eligible.

Exclusion Criteria

1. Caregiver or eligible children have a medical condition that significantly affects diet or eating habits.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Change in Diet quality | baseline and 8 weeks
  Diet quality of the child will be measured by use of an automated self-administered 24-hour dietary recall system (ASA24), completed by the child's caregiver. The ASA24 is a web-based tool that enables automatically coded, self-administered 24-hour diet recalls, providing high-quality dietary data. The ASA24 system is adapted from the United States Department of Agriculture (USDA) Automated Multiple-Pass Method, which has been validated. Validation and evaluation studies of ASA24 have found close agreement with standardized interview-administered 24 hour recall.

SECONDARY OUTCOMES:
Change in Food security - Food Security Survey | baseline and 8 weeks
  Food security status will be assessed using the USDA Food Security Survey. The 18-item USDA Food Security Survey the time period (e.g. last 30 days) and specify lack of resources as the reason for the behavior or experience (e.g. "couldn't afford more food," or "there was not enough money for food") to determine the level food security (very low, low, marginal, and full). Participants are asked to check boxes next to statements that best describe their behavior. These surveys will be administered via REDCap with telephonic support by study staff at baseline and 8 weeks following the initiation of the intervention.
Change in Food security - Hunger Coping Scale | baseline and 8 weeks
  Food security status will be assessed using the Hunger Coping Scale. The five items from the Hunger Coping Scale question the time period (e.g. last 30 days) and specify lack of resources as the reason for the behavior or experience (e.g. "couldn't afford more food," or "there was not enough money for food") to determine the level food security (very low, low, marginal, and full). Participants are asked to check boxes next to statements that best describe their behavior. These surveys will be administered via REDCap with telephonic support by study staff at baseline and 8 weeks following the initiation of the intervention.
Change in Food security - 2-item Nutrition Security Screener (NSS) | baseline and 8 weeks
  Food security status will be assessed using the NSS. These surveys will be administered via REDCap with telephonic support by study staff at baseline and 8 weeks following the initiation of the intervention.
Change in Caregiver diet quality | baseline and 8 weeks
  Caregiver diet quality will be measured by the caregivers completion of the automated self-administered 24-hour dietary recall system (ASA24) for themselves at baseline and 8 weeks following the initiation of the nutrition education intervention. The ASA24, is a web-based tool that enables automatically coded, self-administered 24-hour diet recalls, providing high-quality dietary data. The ASA24 system is adapted from the USDA Automated Multiple-Pass Method, which has been validated.
Change in Caregiver perceived food environment | baseline and 8 weeks
  Perceptions of food environment will be assessed using the Perceived Nutrition Environment Measures survey (NEMS-P). The survey is completed by the person who does the majority of the food shopping in a household to learn about his/her perceptions of the nutrition environments (where food is consumed or purchased, and in the home). Participants are asked to check boxes next to statements that best describe their behavior (e.g. "strongly disagree" to "strongly agree" or "never or rarely" to "almost always". Components within the survey ar examined individually. The survey can discriminate perceptions of nutrition environments between residents of higher- and lower-socioeconomic status (SES) neighborhoods. The NEMS-P will be administered via REDCap with telephonic support by study staff at baseline and 8 weeks following the initiation of the nutrition education intervention.
Change in Caregiver mental health - Loneliness | baseline and 8 weeks
  Caregiver mental health will be measured using the Revised UCLA (R-UCLA) Loneliness Scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item on a scale from "hardly ever" to "often". Minimum score is 3 maximum score is 9; higher scores indicate worse outcome.
Program feasibility - Voucher Redemption | 8 weeks
  Program feasibility will be assessed through voucher redemption
Program feasibility - Home Plate Class Attendance | 8 weeks
  Program feasibility will be assessed through virtual Home Plate class attendance
Program feasibility - Participant Satisfaction | 8 weeks
  Program feasibility will be assessed through participant feedback measured by completion of the participant satisfaction surveys and phone interviews post intervention.
Change in Urine Metabolites | Baseline and 8 weeks
  Urine samples will be collected from subjects at baseline and 8 weeks and measured by metabolomic analysis to quantify association with dietary biomarkers.
Change in Caregiver mental health - Depression | baseline and 8 weeks
  The Center for Epidemiologic Studies Depressive Scale (CES-D) is a 20-item questionnaire that includes a brief self-report for which the scale is designed to measure self-reported symptoms associated with depression experienced in the past week. Participants rate each item on a scale from 0= "Rarely or none of the time (less than 1-day)", 1= "Some or a little of the time (1-2 days)," 2= "Occasionally or a moderate amount of the time (3-4 days," or 3="Most or all of the time (5-7 days)."The scale will be administered via REDCap with telephonic support by study staff at baseline and 8 weeks following the initiation of the interventions. High scores indicating greater depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith LP, Ng SW, Popkin BM. Trends in US home food preparation and consumption: analysis of national nutrition surveys and time use studies from 1965-1966 to 2007-2008. Nutr J. 2013 Apr 11;12:45. doi: 10.1186/1475-2891-12-45. PMID 23577692
- [Background] Zick CD, Stevens RB. Trends in Americans' food-related time use: 1975-2006. Public Health Nutr. 2010 Jul;13(7):1064-72. doi: 10.1017/S1368980009992138. Epub 2009 Nov 30. PMID 19943999
- [Background] Brownell KD. Fast food and obesity in children. Pediatrics. 2004 Jan;113(1 Pt 1):132. doi: 10.1542/peds.113.1.132. No abstract available. PMID 14702462
- [Background] Nelson SA, Corbin MA, Nickols-Richardson SM. A call for culinary skills education in childhood obesity-prevention interventions: current status and peer influences. J Acad Nutr Diet. 2013 Aug;113(8):1031-6. doi: 10.1016/j.jand.2013.05.002. No abstract available. PMID 23885701
- [Background] Kim SA, Moore LV, Galuska D, Wright AP, Harris D, Grummer-Strawn LM, Merlo CL, Nihiser AJ, Rhodes DG; Division of Nutrition, Physical Activity, and Obesity, National Center for Chronic Disease Prevention and Health Promotion, CDC. Vital signs: fruit and vegetable intake among children - United States, 2003-2010. MMWR Morb Mortal Wkly Rep. 2014 Aug 8;63(31):671-6. PMID 25102415
- [Background] Moore LV, Thompson FE. Adults Meeting Fruit and Vegetable Intake Recommendations - United States, 2013. MMWR Morb Mortal Wkly Rep. 2015 Jul 10;64(26):709-13. PMID 26158351
- [Background] Jun S, Thuppal SV, Maulding MK, Eicher-Miller HA, Savaiano DA, Bailey RL. Poor Dietary Guidelines Compliance among Low-Income Women Eligible for Supplemental Nutrition Assistance Program-Education (SNAP-Ed). Nutrients. 2018 Mar 8;10(3):327. doi: 10.3390/nu10030327. PMID 29518042
- [Background] Rivera RL, Maulding MK, Eicher-Miller HA. Effect of Supplemental Nutrition Assistance Program-Education (SNAP-Ed) on food security and dietary outcomes. Nutr Rev. 2019 Dec 1;77(12):903-921. doi: 10.1093/nutrit/nuz013. PMID 31077323
- [Background] Whiteman ED, Chrisinger BW, Hillier A. Diet Quality Over the Monthly Supplemental Nutrition Assistance Program Cycle. Am J Prev Med. 2018 Aug;55(2):205-212. doi: 10.1016/j.amepre.2018.04.027. Epub 2018 Jun 21. PMID 29935945
- [Background] Block JP, Subramanian SV. Moving Beyond "Food Deserts": Reorienting United States Policies to Reduce Disparities in Diet Quality. PLoS Med. 2015 Dec 8;12(12):e1001914. doi: 10.1371/journal.pmed.1001914. eCollection 2015 Dec. PMID 26645285
- [Background] Choi SE, Seligman H, Basu S. Cost Effectiveness of Subsidizing Fruit and Vegetable Purchases Through the Supplemental Nutrition Assistance Program. Am J Prev Med. 2017 May;52(5):e147-e155. doi: 10.1016/j.amepre.2016.12.013. Epub 2017 Jan 30. PMID 28153648
- [Background] Cohen AJ, Richardson CR, Heisler M, Sen A, Murphy EC, Hesterman OB, Davis MM, Zick SM. Increasing Use of a Healthy Food Incentive: A Waiting Room Intervention Among Low-Income Patients. Am J Prev Med. 2017 Feb;52(2):154-162. doi: 10.1016/j.amepre.2016.11.008. PMID 28109458
- [Background] Olsho LE, Klerman JA, Wilde PE, Bartlett S. Financial incentives increase fruit and vegetable intake among Supplemental Nutrition Assistance Program participants: a randomized controlled trial of the USDA Healthy Incentives Pilot. Am J Clin Nutr. 2016 Aug;104(2):423-35. doi: 10.3945/ajcn.115.129320. Epub 2016 Jun 22. PMID 27334234
- [Background] Young CR, Aquilante JL, Solomon S, Colby L, Kawinzi MA, Uy N, Mallya G. Improving fruit and vegetable consumption among low-income customers at farmers markets: Philly Food Bucks, Philadelphia, Pennsylvania, 2011. Prev Chronic Dis. 2013 Oct 3;10:E166. doi: 10.5888/pcd10.120356. PMID 24135390
- [Background] Tester JM, Leung CW, Crawford PB. Revised WIC Food Package and Children's Diet Quality. Pediatrics. 2016 May;137(5):e20153557. doi: 10.1542/peds.2015-3557. Epub 2016 Apr 7. PMID 27244804
- [Background] Parks CA, Stern KL, Fricke HE, Clausen W, Yaroch AL. Healthy Food Incentive Programs: Findings From Food Insecurity Nutrition Incentive Programs Across the United States. Health Promot Pract. 2020 May;21(3):421-429. doi: 10.1177/1524839919898207. Epub 2020 Jan 27. PMID 31984800
- [Background] Marsh DR, Schroeder DG, Dearden KA, Sternin J, Sternin M. The power of positive deviance. BMJ. 2004 Nov 13;329(7475):1177-9. doi: 10.1136/bmj.329.7475.1177. PMID 15539680
- [Background] Gebremedhin S, Baye K, Bekele T, Tharaney M, Asrat Y, Abebe Y, Reta N. Predictors of dietary diversity in children ages 6 to 23 mo in largely food-insecure area of South Wollo, Ethiopia. Nutrition. 2017 Jan;33:163-168. doi: 10.1016/j.nut.2016.06.002. Epub 2016 Jun 16. PMID 27499206
- [Background] Mackintosh UA, Marsh DR, Schroeder DG. Sustained positive deviant child care practices and their effects on child growth in Viet Nam. Food Nutr Bull. 2002 Dec;23(4 Suppl):18-27. PMID 12503228
- [Background] Virudachalam S, Long JA, Harhay MO, Polsky DE, Feudtner C. Prevalence and patterns of cooking dinner at home in the USA: National Health and Nutrition Examination Survey (NHANES) 2007-2008. Public Health Nutr. 2014 May;17(5):1022-30. doi: 10.1017/S1368980013002589. Epub 2013 Oct 10. PMID 24107577
- [Background] Saxe-Custack A, LaChance J, Hanna-Attisha M, Dawson C. Flint Kids Cook: positive influence of a farmers' market cooking and nutrition programme on health-related quality of life of US children in a low-income, urban community. Public Health Nutr. 2021 Apr;24(6):1492-1500. doi: 10.1017/S136898002000395X. Epub 2020 Oct 8. PMID 33028450
- [Background] Kipnis V, Subar AF, Midthune D, Freedman LS, Ballard-Barbash R, Troiano RP, Bingham S, Schoeller DA, Schatzkin A, Carroll RJ. Structure of dietary measurement error: results of the OPEN biomarker study. Am J Epidemiol. 2003 Jul 1;158(1):14-21; discussion 22-6. doi: 10.1093/aje/kwg091. PMID 12835281
- [Background] Moshfegh AJ, Rhodes DG, Baer DJ, Murayi T, Clemens JC, Rumpler WV, Paul DR, Sebastian RS, Kuczynski KJ, Ingwersen LA, Staples RC, Cleveland LE. The US Department of Agriculture Automated Multiple-Pass Method reduces bias in the collection of energy intakes. Am J Clin Nutr. 2008 Aug;88(2):324-32. doi: 10.1093/ajcn/88.2.324. PMID 18689367
- [Background] Kirkpatrick SI, Subar AF, Douglass D, Zimmerman TP, Thompson FE, Kahle LL, George SM, Dodd KW, Potischman N. Performance of the Automated Self-Administered 24-hour Recall relative to a measure of true intakes and to an interviewer-administered 24-h recall. Am J Clin Nutr. 2014 Jul;100(1):233-40. doi: 10.3945/ajcn.114.083238. Epub 2014 Apr 30. PMID 24787491
- [Background] Thompson FE, Dixit-Joshi S, Potischman N, Dodd KW, Kirkpatrick SI, Kushi LH, Alexander GL, Coleman LA, Zimmerman TP, Sundaram ME, Clancy HA, Groesbeck M, Douglass D, George SM, Schap TE, Subar AF. Comparison of Interviewer-Administered and Automated Self-Administered 24-Hour Dietary Recalls in 3 Diverse Integrated Health Systems. Am J Epidemiol. 2015 Jun 15;181(12):970-8. doi: 10.1093/aje/kwu467. Epub 2015 May 10. PMID 25964261
- [Background] Compher CW, Quinn R, Burke F, Piccinin D, Sartor L, Lewis JD, Wu GD. Development of the Penn Healthy Diet screener with reference to adult dietary intake data from the National Health and Nutrition Examination Survey. Nutr J. 2022 Nov 17;21(1):70. doi: 10.1186/s12937-022-00821-w. PMID 36384552
- [Background] Pinard C, Smith TM, Calloway EE, Fricke HE, Bertmann FM, Yaroch AL. Auxiliary measures to assess factors related to food insecurity: Preliminary testing and baseline characteristics of newly designed hunger-coping scales. Prev Med Rep. 2016 Jun 29;4:289-95. doi: 10.1016/j.pmedr.2016.06.021. eCollection 2016 Dec. PMID 27462530
- [Background] Green SH, Glanz K. Development of the Perceived Nutrition Environment Measures Survey. Am J Prev Med. 2015 Jul;49(1):50-61. doi: 10.1016/j.amepre.2015.02.004. PMID 26094227
- [Background] Cosco TD, Prina M, Stubbs B, Wu YT. Reliability and Validity of the Center for Epidemiologic Studies Depression Scale in a Population-Based Cohort of Middle-Aged U.S. Adults. J Nurs Meas. 2017 Dec 1;25(3):476-485. doi: 10.1891/1061-3749.25.3.476. PMID 29268830
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205